CLINICAL TRIAL: NCT04962789
Title: The Impact of Endometrial Compaction on Ongoing Pregnancy Rate in Assisted Reproductive Technology Cycles : Prospective Cohort Study
Brief Title: Endometrial Compaction in Assissted Reproduction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Ahmad Abdelraof Ahmad Askar, assisstant lecturer, Assiut University
Other Study IDs: EC
Record Dates: First submitted 2021-07-10; First posted 2021-07-15 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Infertility, Female
Keywords: infertility; IVF , ICSI; endometrium; compaction
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with compaction: those whose endometrial thickness is calculated to decrease by the time of embryo transfer compared with the thickness at the day of ovulation trigger, analyzed according to the degree of compaction, i.e., 5%, 10%, 15%, or 20% decrease thickness
  Interventions: Diagnostic Test: transvaginal ultrasound on the uterus
- without compaction: those who had an increase in their endometrial thickness or whose thickness decreased less than 5%
  Interventions: Diagnostic Test: transvaginal ultrasound on the uterus

INTERVENTIONS:
Diagnostic Test: transvaginal ultrasound on the uterus — Transvaginal ultrasound measurement to record endometrial thickness 2 times in each cycle:
  In case of fresh cycles: 1)Day of ovulation triggering 2)Day of embryo transfer In case of frozen thawed cycles : 1)End of estrogen phase 2)Day of embryo transfer

SUMMARY:
To record the dynamic change of endometrial thickness (Day of embryo transfer Versus. Day of ovulation trigger administration in case of fresh cycles or end of estrogen phase in frozen cycles), and to investigate the impact of endometrial thickness change on pregnancy outcomes

DETAILED DESCRIPTION:
Clinical pregnancy rate in IVF cycles depends on embryo quality and endometrial receptivity . It is challenging to assess endometrial receptivity. Measuring endometrial thickness by ultrasonography is a simple , noninvasive and accurate method to do so. Many studies have implicated endometrial thickness and pattern as prognostic parameters for successful outcomes in IVF-ET.

Some studies have suggested a minimal thickness for a successful pregnancy to occur, while others have reported adverse effects of increased endometrial thickness above which pregnancy is unlikely to occur.

Now there is a novel hypothesis that not only the initial endometrial thickness can affect implantation rate and clinical pregnancy rate ,but also the decrease in endometrial thickness in the time interval between the ovulation triggering and the embryo transfer or what is called endometrial compaction increases the implantation and clinical pregnancy rate

ELIGIBILITY:
Inclusion Criteria:

* • Infertile women aged 18 years to 40 years undergoing IVF/ ICSI for any indication.

Exclusion Criteria:

* • History of recurrent pregnancy loss (≥ 2 spontaneous abortions) and/or history of recurrent (≥ 2) ICSI failure after embryo transfer.

  * Uterine malformations.
  * Uncorrected hydrosalpinx.
  * Intrauterine conditions affecting pregnancy outcomes such as ( intrauterine adhesions, fibroids, polyps).
  * Any previous hysteroscopic surgery eg. Metroplasty or hysteroscopic myomectomy or uterine surgeries involving the endometrium eg. myomectomy during which uterine cavity was opened.
  * History suggesting endometritis.
  * Use of hCG for endometrial preparation or luteal phase support.
  * Poor quality embryos( according to Istanbul consensus workshop on embryo assessment )

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women undergoing IVF/ICSI.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks after embryo transfer if hCG tested positive
  rate of ongoing pregnancy in patients who have endometrial compaction

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided